CLINICAL TRIAL: NCT00022841
Title: Prevention of Steroid-Induced Osteoporosis in Children
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inadequate eligible subjects to expect sufficient numbers to analyse outcomes.
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23AR002161 (NIH); NIAMS-065
Record Dates: First submitted 2001-08-14; First posted 2001-08-16 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Osteoporosis
Keywords: Bone mineral density (BMD); Children; Glucocorticoids; Osteoporosis; Pediatric; Pamidronate; Steroids
MeSH Terms: conditions — Osteoporosis | interventions — Pamidronate

INTERVENTIONS:
Drug: Pamidronate

SUMMARY:
The purpose of this study is to determine whether the drug pamidronate can safely and effectively improve bone mineral density in growing children who have bone disease caused by taking steroid medications. People who take steroid medications called glucocorticoids, like prednisone or dexamethasone, for long periods almost always have decreased bone density and are at increased risk of breaking a bone. Research has shown that pamidronate improves bone density in adults who take glucocorticoids. However, use of pamidronate is not approved in children because it has not been extensively tested in children. It is possible that children will have a different response or unique problems with the medication because their bones are still growing. We will assign all study participants to one of two groups. One group will receive pamidronate intravenously (through a vein) every 3 months in addition of daily oral calcium and vitamin D and the other group will receive calcium and vitamin D. The study is scheduled to run for 36 months, with visits to the study center once every 3 months.

DETAILED DESCRIPTION:
This is a randomized study to determine whether pamidronate can safely and effectively improve bone mineral density (BMD) in children with glucocorticoid-induced osteoporosis. After we stratify participants on the basis of whether they are taking glucocorticoids for treatment of inflammatory disease or for immunosuppression following organ transplant, we will randomize them to receive daily calcium and vitamin D in addition to 30 mg/kg (1 mg/kg for weight less then 30 kg) of pamidronate in normal saline every 3 months or daily calcium and vitamin D only for 24 months, followed by a 12-month followup period off of therapy. We will measure endpoints at 24 months. The primary endpoint is lumbar spine BMD determined by DEXA. Secondary endpoints will include volumetric BMD of the spine, proximal femur BMD and volumetric BMD, total body bone mineral content (BMC), fracture incidence, bone turnover markers, and growth and skeletal changes. The study radiologist will be blinded to treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Chronic inflammatory disease or transplant recipient, currently on steroid therapy at supraphysiologic dose (greater than hydrocortisone equivalent of 15 mg/m2/day) for more than 6 months
* Bone age less then 14 years in females, 16 years in males, to correspond to < 90% of peak BMD

And

* Presence of glucocorticoid induced bone disease defined by:
* Presence of at least one atraumatic fracture (defined as fracture that occurs during activities of daily living, without a fall), or a vertebral fracture, OR
* AP lumbar spine BMD (determined by DEXA) of more than 2 or more SD below the mean lumbar BMD for a healthy child of similar stature (height age). OR
* A low trauma fracture (suspicious fracture - defined as a fracture the occurs with a fall from standing height or below, and not during a high velocity activity) and AP spine BMD 1.5 or more SD below the mean for height age, OR
* Recent loss of BMD of greater then 3% over a 6 month or greater interval at any one of the following sites, lumbar spine, total hip or whole body (excluding head). OR
* Recent increase in BMD of less then 3% over a 12 month period at all of the three sites listed above.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Lumbar spine BMD determined by DEXA | Measured at Month 24

SECONDARY OUTCOMES:
BMD of the spine, proximal femur BMD and volumetric BMD, total body bone mineral content (BMC), fracture incidence, bone turnover markers, and growth and skeletal changes | Measured at Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca P. Green, MD, PhD, Principal Investigator — Washington University Medical School-St. Louis Children's Hospital
Locations (1):
- Washington University Medical School-St. Louis Children's Hospital, St Louis, Missouri, United States